CLINICAL TRIAL: NCT02198079
Title: A Prospective, Multicenter, Collaborative Study to Determine the Prevalence of Nontuberculous Mycobacteria (NTM) in Pediatric Patients With Cystic Fibrosis in Florida
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: University of Florida (Other)
Responsible Party: Principal Investigator, Andrew Colin, Professor of Pediatrics, University of Miami
Other Study IDs: 20090499
Record Dates: First submitted 2014-02-21; First posted 2014-07-23 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Cystic Fibrosis; Pediatrics
Keywords: non-tuberculous mycobacteria; Pediatrics; Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — one sputum, throat, or bronchoalveolar lavage
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cystic Fibrosis: Children with Cystic Fibrosis
  Interventions: Biological: Sputum

INTERVENTIONS:
Biological: Sputum

SUMMARY:
To determine the prevalence of nontuberculous mycobacterial infection (NTM) in pediatric patients with cystic fibrosis in the State fo Florida. HYPOTHESIS: There is high prevalence of NTM in CF pediatric population in the State of Florida, and likely higher than in the rest of the country.

DETAILED DESCRIPTION:
Non-tuberculous Mycobacteria (NTM) are a heterogeneous group of organisms that have been increasingly reported in North America 1, 2 and recognized to be a pulmonary pathogen in non immunocompromised persons, in middle age-elderly people, non smoking women, apart from the high risk population with underlying lung disease, and also in Cystic fibrosis (CF) population.

Cystic fibrosis (CF) is the most common autosomal recessive disorder in Caucasians, a result of mutations in the Cystic Fibrosis Transmembrane Regulator (CFTR) gene. The carrier rate is estimated at 1:25, and 1:3500 live births in Caucasians are affected with CF. A broadening spectrum of mutations of the CFTR gene has been identified in recent years and a widening array of disorders, particularly of the respiratory system, is expected to be associated with some of these genetic abnormalities. The predisposition to specific airway infections may be a feature of some of these mutations as well as many modifying genes that could alter the course of the disease.

The disease predominantly affects the GI tract and the respiratory system. Infectious complications of the latter are the predominant determinants of morbidity and life expectancy in these patients.

Patients with cystic fibrosis are also at high risk of suffering from chronic airway infections, and one of the increasingly identified microorganisms is non-tuberculous mycobacteria. NTM has been shown to be a potential contributor to the decline in lung function, the major determinant of outcome and longevity of these patients.

Since patients with CF have chronic bacterial pulmonary infections as their disease progresses, the clinical signs and symptoms of NTM are often difficult to distinguish from the underlying disease. Such potential underestimation of the contribution of NTM to the decline of lung function in cystic fibrosis may be an added risk to the eventual outcome of these patients. A variety of microorganisms traditionally considered colonizers of the airways, have been increasing in frequency and assuming new clinical significance5, 6, and previously unknown types of known organisms are taking on a new and ominous clinical significance.7 To the practicing clinician NTM appears to be increasing in incidence among the CF population, but the significance of this observation has not been firmly established. The concept of "colonization," defined as the isolation of the organism from the respiratory tract without evidence of tissue invasion, was supported by several investigators in the past, mainly in association with M. avium-complex infection.8, 9 With the emergence of high resolution CT scanning (HRCT), it now appears that many of these patients have features of parenchymal involvement, usually of a nodular pattern, suggesting that the term "colonization," at least in some patients, may be erroneous10, this notion has also been supported by direct bioptic evidence11, indicating the possibility that the full significance of infection with NTM may be underappreciated in patients with CF. It has been proposed that rather than using terminologies such as colonization and active disease, the distinction should be between patients who require immediate therapy on the basis of the rapid progression of their disease and those in whom the decision can be delayed.12 The repeated isolation of the same Mycobacterium from a patient with CF may be indicative of indolent infection and these patients may be at risk of developing clinical symptoms that will ultimately require treatment. This observation is supported by a series of autoptic studies13 indicating that patients with CF who have multiple positive sputum cultures for NTM are more likely to have histologic evidence of granulomatous mycobacterial disease. An additional study11 reports of a patient who had bioptic evidence of granulomas with NTM infection resulting in fulminant disease some 14 years later, suggesting that frank infections may be subclinical for a long period of time. The predictable but variable progression of the lung disease inherent to CF cannot be easily uncoupled from a possible contribution that chronic infection with NTM may add to the slope of such decline. Thus the role of such silent infections in exacerbating the decline of pulmonary function in such patients remains to be elucidated. From the clinical perspective subtle changes on serial high resolution computerized tomography of the chest (HRCT) may enable earlier diagnosis and intervention prior to the development of cavitation and/or irreversible lung damage.10 Of the NTM, Mycobacterium abscessus is a member of the rapidly growing mycobacteria. With improvements in identification, it is now known that this organism accounts for approximately 80% of rapidly-growing mycobacterial respiratory disease isolates.9 Prior to the 1990s, there were few reports of clinically important NTM infection complicating CF of which seven were cases of M. abscessus.11 Although the natural history of this disease can vary, it appears to follow a more fulminant course in patients with underlying lung diseases such as cystic fibrosis.14 The treatment of M. abscessus is complex. The isolates are uniformly resistant to standard antituberculosis drugs and are generally susceptible only to parenteral antibiotics and the newer oral macrolides. The organism is notoriously difficult to eradicate. In a report of 154 patients infected with rapidly growing mycobacteria14, only 10 patients infected with M. abscessus exhibited a "cure," the latter being defined as a return of respiratory symptoms to baseline and reversion of sputum to smear and culture negativity for at least 1 year. It has been noted for many years that the rates of infection and morbidity with and from NTM in non-CF patients have been increasing.1, 9 This notion has been recently supported by a report on the prevalence of mycobacterial infection in Ontario. The prevalence rose significantly (p<0.001) from 9.1/100,000 in 1997 to 16.5/100,000 in 2002, and 14.2/100,000 in 2003. A coincidental significant (<0.001) decline in the rate of M. tuberculosis infection from 6.9/100,000 in 1997 to 5.4/100,00 in 2003 was noted15. Whether such a trend of increasing prevalence of NTM also occurs in CF has not been formally addressed in the literature.

A number of studies from the US and Europe addressing the epidemiology of NTM in cystic fibrosis has been published. These studies suggest a large variability in the incidence and the nature of the infecting organisms between various regions of the world, and various institutions. While the clinical impression would support a trend of increasing prevalence of NTM in CF parallel to non-CF patients, the absence of repeated studies and the limitations imposed by the inconsistencies amongst centers and regions, does not allow a firm statement on this subject.

The increasing rates of infection and morbidity from NTM in non-CF patients 1, 2 is likely similarly trending amongst patients with CF. In the US, a 1992 study from the University of North Carolina at Chapel Hill 3 revealed a high prevalence of CF patients with NTM infection in the southeastern United States. Of 87 patients studied 17 (19.5%) had at least one positive culture for NTM. A 1993 study was reported from the University of Washington 4 revealing a prevalence of 12.5% amongst their 64 adult patients.

The key publications on prevalence of NTM in patients with CF in the US by Olivier et al5 revealed an overall prevalence of 13%, with the most common organisms in adults being M. avium- complex (MAC).

Data on the prevalence and significance of NTM infections in younger patients with CF are less clear. Several studies suggest that NTM infection in CF pediatric population is low 3-7 but the numbers vary around the globe. A study from Necker Hospital for Sick Children in Paris8 revealed a prevalence of 5 % in children with a mean age of age 11.9 y o (2.5 to 22 y o). It also revealed that M. abscessus was the prevailing organism among the pediatric population, rather than MAC, the commonest organism in adults.

The Olivier studies 5 confirmed that the prevalence of NTM is particularly high in the southeastern USA, as previously suggested by a study from the adult CF center of the University of North Carolina at Chapel Hill 3 that revealed a prevalence of 19.5%. It is therefore of particular interest that a recent pediatric study from the same medical center 9 retrospectively reviewed CF patients younger than 12 years old and found 6.1% overall prevalence of NTM in BALs over 3 years, and 3.9 % using medical record examination over a 10- year period.

This information that is collected will help to deepen the understanding of the nature of the microbiology of our CF pediatric population, and to what extent NTM play a role in the colonization and possible disease causation in this region of the country. The investigators think this role is underestimated. Once the information becomes available, The investigators will be able to make better plans of dealing with this infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have a diagnosis of Cystic Fibrosis and are 18 or below years of age

Exclusion Criteria:

* Patients that are above 18 years of age and or patients that do not have the diagnosis of Cystic fibrosis

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Cystic Fibrosis aged from 0 to 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2010-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Positive culture for non-tuberculous mycobacteria (NTM) | At visit one
  Sputum or bronchoalveolar lavage sample will be analyzed for culture of NTM

SECONDARY OUTCOMES:
Prevalence of NTM | Week 52
  The prevalence of the NTM found in the cultures will be determined from this sample

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Colin, MD, SM, Principal Investigator — University of Miami; Shatha Yousef, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miller School of Medicine, Miami, Florida, United States